CLINICAL TRIAL: NCT06318884
Title: A Phase Ia/Ib Dose-escalation and Dose-expansion Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of SCTB35 in Patients With CD20+ Relapse/Refractory B-cell Non-Hodgkin Lymphoma
Brief Title: A First-in-human Study of SCTB35 in Patients With Relapse/Refractory B-cell Non-Hodgkin Lymphoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCTB35-X101
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Non-Hodgkin Lymphoma, B-cell
Keywords: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCTB35 (Experimental): SCTB35 injection is subcutaneously given every week for the first 4 cycles, and thereafter every 3 weeks. Cycles will be repeated every 3 weeks until disease progression, study discontinuation, or death, whichever occurs first.
  Interventions: Drug: SCTB35 injection

INTERVENTIONS:
Drug: SCTB35 injection — SCTB35 will be subcutaneously administered at a dose as specified in the respective dose-escalation cohorts. Then, the RP2D and another appropriate dose of SCTB35 will be applied for the dose-expansion cohorts.
  Other Names: none other names

SUMMARY:
This is a Phase I clinical study designed to evaluate the safety, tolerability, and pharmacokinetics, and preliminary efficacy of SCTB35 monotherapy, an bispecific antibody, in patients with relapsed and/or refractory B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
This is the first-in-human study of SCTB35, containing the dose-escalation and dose-expansion parts. The escalation cohorts will be enrolled to explore the maximum tolerated dose and recommended phase II dose (RP2D). A Safety Monitoring Committee (SMC) will review the accumulated safety data and other available data, and make a recommendation to each dose level of SCTB35 in the escalation cohorts. The expansion cohorts will be initiated after the RP2D is confirmed, and to further compare the preliminary efficacy and safety of SCTB35 at two dose levels that appropriately recommended by SMC.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if all the following conditions are met:

1. Age ≥ 18 years
2. Histologically or cytologically confirmed CD20+ mature B-cell neoplasm

   For dose-escalation phase:
   1. De novo or transformed diffuse large B-cell lymphoma (DLBCL)
   2. High-grade B-cell lymphoma (HGBCL)
   3. Primary mediastinal large B-cell lymphoma (PMBCL)
   4. Follicular lymphoma (FL)
   5. Mantle cell lymphoma
   6. Small lymphocytic lymphoma (SLL)
   7. Marginal zone lymphoma (MZL) (nodal, extranodal or mucosa associated)

   For dose expansion phase:
   1. FL cohort: histologic confirmed FL grade 1, 2, or 3a at initial diagnosis without clinical or pathological evidence of transformation
   2. LBCL cohort: including histologic confirmed DLBCL, not otherwise specified (NOS), Epstein-Barr virus+ DLBCL, transformed DLBCL from indolent subtypes, HGBCL, NOS, double/triple-hit HGBCL, FL grade 3b, and PMBCL
3. For dose-escalation phase:

   Relapsed, progressive and/or refractory disease after adequate systemic therapy containing at least an anti-CD20 monoclonal antibody (e.g. rituximab)
   1. Patients must have exhausted or are ineligible for all standard therapeutic options
   2. Patients with indolent lymphoma (FL, MZL or SLL) must have a need for treatment initiation based on symptoms and/or disease burden

   For dose-expansion phase:

   Relapsed, progressive and/or refractory disease following ≥ 2 prior lines of adequate systemic therapy containing at least an anti-CD20 monoclonal antibody (e.g. rituximab)
4. At least 1 measurable site of disease based on computed tomography (CT) or magnetic resonance imaging (MRI) (defined as a clearly nodal lesion with the long axis > 1.5 cm or extranodal lesion with the long axis > 1.0 cm). Lesions that have previously received radiotherapy can be considered measurable only after confirming the presence of progression or residual lesions. (for the dose-escalation phase: a evaluable site of disease is allowed).
5. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
6. Adequate hepatic/hematologic/renal/cardiac functions indicated by laboratory values

   1. Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L within 7 days before first dose of study drug (without growth factor support). There is an exception for patients with bone marrow involvement in which case ANC must be ≥ 0.75 x 10^9/L
   2. Platelets > 75 x 10^9/L within 7 days before first dose of study drug (without growth factor support or transfusion). There is an exception for patients with bone marrow involvement in which case platelets must be ≥ 50 x 10^9/L
   3. Hemoglobin > 90 g/L within 7 days before first dose of study drug (independent of growth factor support or transfusion).
   4. Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or creatinine clearance ≥ 45 mL/min as estimated by Cockcroft-Gault equation
   5. Adequate liver function indicated by: i) Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase ≤ 3 x ULN; ii) Alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase ≤ 3 x ULN; iii) Total bilirubin level ≤ 1.5 x ULN (unless documented Gilbert's syndrome).
   6. Left ventricular ejection fraction ≥ 50%;
7. Expected survival time is more than 3 months

Exclusion Criteria:

A patient who conforms to any of the following criteria should be excluded from the study:

1. Any prior therapy with an bispecific antibody of the same class
2. Eligible for high dose chemotherapy with hematopoietic stem cell transplantation (HSCT)
3. Known central nervous system (CNS) involvement by lymphoma
4. Known past or current malignancy other than inclusion diagnosis, with the following exceptions:

   1. Cervical carcinoma of Stage Ib or less
   2. Non-invasive basal cell or squamous cell skin carcinoma
   3. Non-invasive, superficial bladder cancer
   4. Prostate cancer with a current prostate-specific antigen (PSA) level <0.1 ng/mL
   5. Any curable cancer with a complete response (CR) of >2 years duration
5. Known clinically significant cardiac disease, including:

   1. Onset of unstable angina pectoris or acute myocardial infarction within 6 months prior to signing Informed Consent Form (ICF)
   2. Congestive heart failure prior to signing ICF (meets the criteria of New York Heart Association Classification III or IV)
   3. Clinically significant arrhythmia prior to signing ICF
6. History of interstitial lung disease or uncontrolled lung diseases, or evidence of dyspnea at rest or pulse oximetry < 93% while breathing room air.
7. Confirmed history or current autoimmune disease or other diseases resulting in permanent immunosuppression or requiring permanent immunosuppressive therapy (including >20mg/day prednisolone [or equivalent], but low-dose prednisolone is allowed). The well controlled autoimmune disease can be enrolled at investigator's discretion, including:

   1. Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone
   2. Patients with a history of type 1 diabetes mellitus who were well controlled (defined as a screening hemoglobin A1c < 8% and no urinary ketoacidosis)
   3. Patients with skin disease who were not treated with systemic corticosteroid
8. History of seizure disorder or confirmed progressive multifocal leukoencephalopathy (PML)
9. History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
10. Known any major episode of active infection requiring treatment with systemic antibiotics within 2 weeks prior to signing ICF
11. Positive for human immunodeficiency virus (HIV) antibody. Positive for hepatitis B antibody (except for only the positive HBsAb) with detectable hepatitis B virus (HBV) DNA. Positive for hepatitis C antibody with detectable hepatitis C virus (HCV) RNA
12. Chimeric antigen receptor T-cell (CAR-T) therapy within 100 days prior to first SCTB35 administration (only applicable for dose-expansion phase)
13. Autologous HSCT within 100 days prior to first SCTB35 administration, or any prior allogeneic HSCT or solid organ transplantation
14. Received major surgery within 4 weeks prior to first SCTB35 administration, or planned to receive major surgery during the study
15. Received any chemotherapeutic agent, other anti-cancer agent, or investigational drug (monoclonal antibody, radioimmunoconjugate, antibody-drug conjugate or otherwise) within 4 weeks or five half-lives of the drug, whichever is shorter, prior to first SCTB35 administration
16. Exposed to live or live attenuated vaccine within 4 weeks prior to first SCTB35 administration, or planned to receive these vaccines during the study
17. Pregnancy or breast feeding. During the study and for 6 months after last administration of SCTB35, a woman of childbearing potential or a man who is sexually active with a woman of childbearing potential disagrees to practice a highly effective method of birth control.
18. Patient has any condition for that, in the opinion of the investigator, participation could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dose-escalation part: dose limited toxicity (DLT) | During the first cycle (21 days)
  To determine the maximum tolerated dose (MTD) and/or RP2D to be studied in the dose-expansion part
Dose-escalation part: incidence rate of adverse event (AE) | From first dose until 28 days after last dose of study drug or until study completion or participant withdrawal (up to 3 years)
  To evaluate the incidence rates of treatment emergent adverse event (TEAE), treatment-related TEAE (TRAE), serious adverse event (SAE), adverse event with special interest (AESI)
Dose-expansion part: objective response rate (ORR) | From first dose until up to 2 years
  ORR is defined as the percentage of patients achieving complete response (CR) or partial response (PR) as determined by the investigator according to the Lugano Criteria 2014

SECONDARY OUTCOMES:
Dose-escalation part: ORR | From first dose until up to 2 years
  ORR is defined as the percentage of patients achieving CR or PR as determined by the investigator according to the Lugano Criteria 2014
Dose-escalation part: CR rate (CRR) | From first dose until up to 2 years
  CR rate is defined as the percentage of patients with CR as determined by the investigator according to the Lugano Criteria 2014
Dose-escalation part: best of overall response (BOR) | From first dose until up to 2 years
  BOR is defined as the percentage of patients achieving best response from the first dose to first documented disease progression (PD) or new anticancer therapy, whichever occurs first, as determined by the investigator according to the Lugano Criteria 2014
Dose-escalation part: duration of response (DOR) | From first dose until up to 2 years
  DOR is defined as the time from first documented objective response to PD or death due to any cause, whichever occurs first, as determined by the investigator according to the Lugano Criteria 2014
Dose-escalation part: progression-free survival (PFS) | From first dose until up to 2 years
  PFS is defined as the time from first dose to first documented PD or death due to any cause, whichever occurs first, as determined by the investigator according to the Lugano Criteria 2014
Dose-escalation part: time to response (TTR) | From first dose until up to 2 years
  TTR is defined as the time from first dose to first documented objective response observed for patients who achieved a CR or PR, as determined by the investigator according to the Lugano Criteria 2014
Dose-escalation part: overall survival (OS) | From first dose until up to 5 years
  OS is defined as the time from first dose to death due to any cause
Dose-escalation part: blood concentrations of SCTB35 | From first dose until up to 2 years
  The pharmacokinetics of SCTB35 will be analyzed based on the drug concentrations at respective timepoints in the blood samples (or blood derivative)
Dose-escalation part: anti-drug antibodies of SCTB35 | From first dose until up to 2 years
  Blood samples (or blood derivative) will be screened for antibodies binding to SCTB35
Dose-expansion part: CRR | From first dose until up to 2 years
  CR rate is defined as the percentage of patients with CR as determined by the investigator according to the Lugano Criteria 2014
Dose-expansion part: BOR | From first dose until up to 2 years
  BOR is defined as the percentage of patients achieving best response from the first dose to first documented PD or new anticancer therapy, whichever occurs first, as determined by the investigator according to the Lugano Criteria 2014
Dose-expansion part: DOR | From first dose until up to 2 years
  DOR is defined as the time from first documented objective response to PD or death due to any cause, whichever occurs first, as determined by the investigator according to the Lugano Criteria 2014
Dose-expansion part: PFS | From first dose until up to 2 years
  PFS is defined as the time from first dose to first documented PD or death due to any cause, whichever occurs first, as determined by the investigator according to the Lugano Criteria 2014
Dose-expansion part: TTR | From first dose until up to 2 years
  TTR is defined as the time from first dose to first documented objective response observed for patients who achieved a CR or PR, as determined by the investigator according to the Lugano Criteria 2014
Dose-expansion part: OS | From first dose until up to 5 years
  OS is defined as the time from first dose to death due to any cause
Dose-expansion part: AE | From first dose until up to 2 years
  To evaluate the incidence rates of TEAE, TRAE, SAE, AESI
Dose-expansion part: blood concentrations of SCTB35 | From first dose until up to 2 years
  The pharmacokinetics of SCTB35 will be analyzed based on the drug concentrations at respective timepoints in the blood samples (or blood derivative)
Dose-expansion part: anti-drug antibodies of SCTB35 | From first dose until up to 2 years
  Blood samples (or blood derivative) will be screened for antibodies binding to SCTB35

CONTACTS AND LOCATIONS:
Overall Officials: Yuqin Song, M.D., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (3):
- China (3):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality